CLINICAL TRIAL: NCT01082926
Title: Phase I Study of Cellular Immunotherapy for Recurrent/Refractory Malignant Glioma Using Intratumoral Infusions of GRm13Z40-2, An Allogeneic CD8+ Cytolitic T-Cell Line Genetically Modified to Express the IL 13-Zetakine and HyTK and to be Resistant to Glucocorticoids, in Combination With Interleukin-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07082; NCI-2010-00303
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Ependymoma; Anaplastic Meningioma; Anaplastic Oligodendroglioma; Brain Stem Glioma; Ependymoblastoma; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Grade III Meningioma; Meningeal Hemangiopericytoma; Mixed Glioma; Pineal Gland Astrocytoma; Brain Tumor
Keywords: adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic meningioma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult ependymoblastoma; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult grade III meningioma; adult meningeal hemangiopericytoma; adult mixed glioma; adult pineal gland astrocytoma; recurrent adult brain tumor; Los Angeles
MeSH Terms: conditions — Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — aldesleukin; Interleukin-2; Interleukins; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive intratumoral GRm13Z40-2 therapeutic allogeneic lymphocytes over 10 minutes on days 1 and 3 and intratumoral aldesleukin over 3 hours on days 2-5 (days 1-5 in week 2). Treatment repeats every week for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: therapeutic allogeneic lymphocytes; Biological: aldesleukin; Other: laboratory biomarker analysis; Procedure: positron emission tomography

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Given intratumorally
  Other Names: ALLOLYMPH
Biological: aldesleukin — Given intratumorally
  Other Names: IL-2; interleukin II; Proleukin; recombinant human interleukin-2; recombinant interleukin-2; TCGF, interleukin
Other: laboratory biomarker analysis — Optional correlative studies
Procedure: positron emission tomography — Optional correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
RATIONALE: Biological therapies, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop tumor cells from growing. Donor T cells that are treated in the laboratory may be effective treatment for malignant glioma. Aldesleukin may stimulate the white blood cells to kill tumor cells. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best way to give therapeutic donor lymphocytes together with aldesleukin in treating patients with stage III or stage IV malignant glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of GRm13Z40-2 CTL CNS loco-regional cellular immunotherapy in research participants with recurrent or refractory/ progressive malignant glioma (WHO Grades 3 or 4).

II. To assess the safety of convection enhanced delivery (CED) of recombinant human Interleukin-2 (rhuIL-2) used in conjunction with GRm13Z40-2 CTL adoptive transfer.

SECONDARY OBJECTIVES:

I. To investigate the ability of 9-(4-fluoro-3-hydroxy-methyl-butyl) guanine (18FHBG) positron emission tomography PET to image GRm13Z40-2 CTL's in research participants.

II. To study the impact of concurrent dexamethasone administration on the tempo and magnitude of T cell allograft rejection responses in treated research participants by tracking the frequency of anti-GRm13Z40-2 immune responses in serially acquired peripheral blood samples.

III. To evaluate ganciclovir administration for ablating transferred GRm13Z40-2 in vivo should significant graft-mediated toxicities be encountered.

OUTLINE: Patients receive GRm13Z40-2 therapeutic allogeneic lymphocytes intratumorally (IT) over 10 minutes on days 1 and 3 and aldesleukin IT over 3 hours on days 2-5 (days 1-5 in week 2). Treatment repeats every week for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed annually for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological verification of grade III or IV MG at original diagnosis
* Radiographic evidence of progression/recurrence of the measurable disease more than 12 weeks after the end of radiation therapy
* Expression of IL13Ralpha2 by immunohistochemistry
* Karnofsky performance status (KPS) >= 60
* Disease recurrence/progression in the cerebral hemisphere, which is in at least one area of enhancement amenable to biopsy after protocol enrollment in the following locations:

  * Adjacent or near previous resection cavity
  * Distant from primary location; this includes tumor spread to contralateral hemisphere, corpus callosum, thalamus, basal ganglion, or subependymal locations
* Research participant has recovered from toxicity of prior therapies; an interval of at least 12 weeks must have elapsed since the completion of radiation therapy; at least 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen; and at least 4 weeks since the completion of a non-nitrosourea-containing cytotoxic chemotherapy regimen; if a patient's most recent treatment was with a targeted agent only, and s/he has recovered from any toxicity of this targeted agent, then a waiting period of only 2 weeks is needed from the last dose and the start of study treatment, with the exception of bevacizumab where a wash out period of at least 4 weeks is required before starting study treatment
* History of prior treatment with Temodar if no evidence of intolerance; documentation of intolerance to Temodar is not required
* Creatinine < 1.6
* White blood cell (WBC) >= 2,000/dl (or absolute neutrophil count [ANC] > 1,000) Platelets >= 100,000/dl unsupported by transfusion or growth factor, international normalized ratio (INR) < 1.3
* Bilirubin < 1.5
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 2 X upper limits of normal
* Female research participants of childbearing potential must not be pregnant as evidenced by a serum beta-HCG pregnancy test obtained within 7 days of enrollment
* Research participants having reproductive potential must agree to use effective contraception during participation on this protocol
* In the opinion of the neurosurgeon, research participant requires on-going dexamethasone therapy

Exclusion Criteria:

* Survival expectation less than 4 weeks
* Pulmonary- Requirement for supplemental oxygen use that is not expected to resolve within 2 weeks, Cardiac- Uncontrolled cardiac arrhythmia, hypotension requiring pressor support, Renal- Dialysis dependent, Neurologic- refractory seizure disorder, clinically evident progressive encephalopathy
* Tumors with the following characteristics:

  * Large tumor recurrence causing significant symptoms from brain shift or mass effect, and thus not requiring "decompressive" craniotomy
  * Tumors located primarily in the basal ganglion or thalamus
  * Tumors with significant involvement of midbrain, cerebellum, pons and medulla will be excluded due to neurological risks associated with edema exacerbation from therapy
* Research participants with any non-malignant intercurrent illness which is either poorly controlled with currently available treatment, or which is of such severity that the investigators deem it unwise to enter the research participant on protocol shall be ineligible
* Positive human immunodeficiency virus (HIV) serology based on testing within 4 weeks of enrollment
* Research participants being treated for severe infection or who are recovering from major surgery are ineligible until recovery is deemed complete by the investigator
* Failure to understand the basic elements of the protocol and/or the risks/benefits of participating in this pilot study
* History of ganciclovir and/or magnetic resonance imaging (MRI) contrast allergy or intolerance History of intolerance to IL-2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety of GRm13Z40-2 CTL CNS loco-regional cellular immunotherapy | Daily for first 2 weeks, weekly for month 1, every other week for month 2 , monthly for 6 months
Safety of convection enhanced delivery (CED) of recombinant human Interleukin-2 (rhuIL-2) used in conjunction with GRm13Z40-2 CTL adoptive transfer | Weeks 1 and 2
Toxicity as assessed by NCI CTCAE version 4.0 | During treatment and up to 21 days after the last GRm13Z40-2 or CED rhuIL-2 infusion

SECONDARY OUTCOMES:
Ability of 9-(4-fluoro-3-hydroxy-methyl-butyl) guanine (18FHBG) positron emission tomography PET to image GRm13Z40-2 CTLs | Prior to immunotherapy and 3 weeks post immunotherapy
Impact of concurrent dexamethasone on the tempo and magnitude of T cell allograft rejection responses by tracking the frequency of anti-GRm13Z40-2 immune responses in serially acquired peripheral blood samples | Post infusion day 1, weeks 2-4 and week 8
Evaluation of ganciclovir administration for ablating transferred GRm13Z40-2 in vivo should significant graft-mediated toxicities be encountered | When/if grade 3 or 4 toxicity occurs

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Badie, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States